CLINICAL TRIAL: NCT04524728
Title: Patterns of Treatment and Outcome of Palbociclib Plus Endocrine Therapy in Hormone Receptor-positive (HR+)/HER2 Receptor-negative (HER2-) Metastatic Breast Cancer (MBC): a Real World Multicentre Italian Study
Brief Title: Patterns of Treatment and Outcome of Palbociclib Plus Endocrine Therapy
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: CE 2295
Record Dates: First submitted 2020-07-09; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-07

CONDITIONS: Breast; Neoplasm Malignant; Female
Keywords: endocrine therapy; metastatic breast cancer; palbociclib; real world; visceral involvement
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — palbociclib; Letrozole; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: Patients that received palbociclib combined with letrozole 2.5 mg
  Interventions: Drug: Palbociclib; Drug: Letrozole 2.5mg
- Cohort B: Patients that received palbociclib combined with fulvestrant 500 mg
  Interventions: Drug: Palbociclib; Drug: Fulvestrant

INTERVENTIONS:
Drug: Palbociclib — tablets
  Other Names: ibrance
Drug: Letrozole 2.5mg — tablets
  Other Names: Femara
  Groups: Cohort A
Drug: Fulvestrant — intramuscolar injections
  Other Names: Faslodex
  Groups: Cohort B

SUMMARY:
This is a multicentre real-world experience aimed at verifying the outcome of palbociclib plus ET in an unselected population of MBC patients. The primary endpoint is the clinical benefit rate (CBR); secondary aims are the median PFS (mPFS), overall survival (OS) and safety.

DETAILED DESCRIPTION:
This is an open-label, longitudinal, prospective, multicentre cohort study. Eligible patients are pre- and postmenopausal women with a histologically proven HR+ MBC, candidate to receive palbociclib plus endocrine therapy (ET) as first or subsequent line of therapy according to their contingent clinical situation. Additional inclusion criteria are HER2- disease (immunohistochemistry (IHC) 0-1+ or IHC 2+, confirmed as fluorescence in situ hybridization [FISH] negative), presence of measurable or evaluable lesions and life expectancy of at least 4 months. They need to have adequate bone marrow, hepatic and renal function, according to clinical practice guidelines for antineoplastic drug administration. Previous chemotherapy or ET for metastatic disease is allowed. Patients receive palbociclib 125 mg daily, 3 weeks on/1 week off in a 28-day cycle, combined with letrozole 2.5 mg administered orally on a continuous daily dosing schedule (cohort A) or fulvestrant at the dose of 500 mg intramuscular on days 1, 14, 28, then every 4 weeks thereafter (cohort B). Premenopausal women receive a GnRH analogue in combination with ET and palbociclib. Treatment is administered until documented disease progression (PD), unacceptable toxicity or patient refusal. The tumour assessment is performed approximately every 16 weeks. Treatment efficacy is evaluated by Response Evaluation Criteria In Solid Tumors (RECIST version 1.1). A complete blood count and organ function test is performed before each cycle, through study completion, an avarange of 1 year. No pre-specified treatment modifications are planned; dose reductions, delay or discontinuations of palbociclib are performed according to observed side effects. AEs are recorded and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) (version 5.0).

The primary aim of the study is to analyse the activity of palbociclib plus ET in terms of clinical benefit rate that is defined as the percentage of patients experiencing complete response (CR), partial response (PR), or stable disease (SD) lasting 6 months or more. Secondary aims include the evaluation of the safety of the treatments, progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Pre- and postmenopausal women with a histologically proven HR+MBC, candidate to receive palbociclib plus ET as first or subsequent line of therapy according to their contingent clinical situation.
* HER2- disease (IHC 0-1 or IHC 2, confirmed as FISH negative), presence of measurable or evaluable lesions and life expectancy of at least 4 months.
* Adequate bone marrow, hepatic and renal function, according to clinical practice guidelines for antineoplastic drug administration

Exclusion Criteria:

* ER- PgR- disease
* HER2+ disease (IHC 3 or IHC 2, confirmed as FISH positive)
* Any cardiovascular, renal or hepatic condition that would compromise conditions in the opinion of the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred-ninety-one patients (92 in cohort A, 99 in cohort B) were enrolled and treated and 182 were evaluable for the analysis. Median age was 62 years (range 47-79)
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Clinical Benefit Rate (CBR) | From the date of randomization through study completion, assessed up to 16 weeks
  the percentage of patients experiencing complete response (CR), partial response (PR), or stable disease (SD) lasting 6 months or more

SECONDARY OUTCOMES:
Median PFS | From date of randomization until the date of first documented progression, assessed up to 16 weeks through study completion
  the time interval from the start of therapy with palbociclib plus ET to the date of
Overall survival | from the date of randomization until the date of death from any cause or lost of follow-up, whichever came first, assessed up to 100 months.
  the interval from therapy start to the date of death or of last follow-up evaluation
Drug safety and tolerability | at day 1 of any cycle from the date of the start of therapy through study completion, an avarange of 1 year
  Incidence of Treatment-emergent adverse events (safety and tolerability) using CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella Palumbo, MD, PhD, Principal Investigator — ICS Maugeri, IRCCS, Department of Medical Oncology, Pavia, italy
Locations (1):
- Istituti Clinici Scientifici Maugeri IRCCS, Pavia, Italy